CLINICAL TRIAL: NCT07083258
Title: The Effect of Inspiratory Muscle Training on Respiratory Parameters, Balance, Trunk Endurance and Trunk Isokinetic Muscle Strength in Elite Freestyle Female Wrestling Athletes
Brief Title: The Effect of Inspiratory Muscle Training on Respiratory Parameters, Balance, Trunk Endurance and Trunk Isokinetic Muscle Strength in Wrestling Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, MİNE PEKESEN KURTÇA, Ass.Prof., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMÜ2025/257
Record Dates: First submitted 2025-07-02; First posted 2025-07-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Physiological Performance in Healthy Female Athletes
Keywords: Inspiratory Muscle Training; Elite Athletes; Female Wrestlers; Trunk Muscle Endurance; Balance; Cardiopulmonary Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training Program (Experimental): Participants in this group will receive a progressive inspiratory muscle training (IMT) program using the POWERbreathe Plus device. Training will be conducted 5 days per week for 4 weeks. The intensity will start at 50% of the participant's measured maximal inspiratory pressure (MIP) and will be increased by 10% each week, reaching 80% in the final week. All training will be performed in addition to the athletes' regular wrestling sessions. Participants in this group will be assessed for respiratory parameters, trunk endurance, balance, and trunk isokinetic muscle strength before and after the intervention.
  Interventions: Device: Progressive Inspiratory Muscle Training (IMT)
- Control Group (Placebo Comparator): Participants in the control group will receive a sham inspiratory muscle training program using the same device. The training intensity will be fixed at 15% of the initial MIP throughout the 4-week period to produce a placebo effect. The frequency and duration of training will mirror that of the experimental group. Participants will undergo identical pre- and post-intervention evaluations.
  Interventions: Other: Placebo Training

INTERVENTIONS:
Device: Progressive Inspiratory Muscle Training (IMT) — The intervention involves the application of inspiratory muscle training using the POWERbreathe Plus device. Training will be conducted at an initial intensity of 50% of the individual's MIP and will be increased weekly by 10%, reaching 80% by week four. Sessions will take place 5 days per week and consist of 2 sets of 30 repetitions per day, with 2-minute rest intervals between sets. This training aims to improve inspiratory muscle strength and endurance, as well as core stability, respiratory function, dynamic balance, and trunk isokinetic strength.
  Arms: Inspiratory Muscle Training Program
Other: Placebo Training — The placebo group will perform identical training sessions using the same device but with a constant minimal resistance set at 15% of the initial MIP, insufficient to induce a physiological training effect. This intervention is designed to control for placebo response. Assessment protocols will be identical to those in the experimental group.
  Arms: Control Group

SUMMARY:
Title:

The Effects of Inspiratory Muscle Training on Respiratory Parameters, Balance, Trunk Endurance, and Trunk Isokinetic Muscle Strength in Elite Female Freestyle Wrestlers

Objective:

This experimental study aims to investigate the effects of inspiratory muscle training on respiratory functions, trunk muscle strength, endurance, and balance in elite female freestyle wrestlers.

Methods:

This randomized controlled trial will include 30 elite female freestyle wrestlers aged between 16 and 22. Participants will be randomly assigned to either an intervention group or a placebo control group using a simple randomization method. The intervention group will receive progressive inspiratory muscle training with the POWERbreathe Plus device, 5 days per week for 4 weeks. The training load will increase weekly. The control group will undergo low-resistance inspiratory training set at 15% of their baseline maximal inspiratory pressure (MIP), serving as a placebo. Pre- and post-intervention assessments will be conducted by a blinded evaluator.

DETAILED DESCRIPTION:
This study aims to investigate the multifaceted effects of inspiratory muscle training (IMT) on performance parameters in elite female freestyle wrestlers within the field of cardiopulmonary physiotherapy and rehabilitation. Unlike most studies in the sports physiotherapy literature, this research goes beyond respiratory parameters to include key functional outcomes such as balance, trunk endurance, and isokinetic trunk muscle strength.

Scientific Background and Rationale Freestyle wrestling is a physically demanding sport that requires simultaneous, dynamic use of both upper and lower extremities, along with high levels of strength, balance, and coordination. Success in competition is closely linked to factors such as postural stability, core muscle activation, and the ability to generate isometric and dynamic force. However, the contribution of respiratory muscles to athletic performance has often been overlooked or assessed only indirectly in previous studies.

Given the high-intensity and short-duration nature of wrestling matches, increased ventilatory demand places a significant burden on the diaphragm and accessory respiratory muscles. Recent evidence suggests that IMT not only improves pulmonary function but also enhances core stabilization and postural control. Therefore, directly assessing the effects of IMT on respiratory and trunk muscle performance in elite female wrestlers addresses a notable gap in the literature.

Study Design This is a randomized controlled experimental study involving 30 elite female freestyle wrestlers affiliated with the Turkish Olympic Preparation Center (TOHM-Trabzon). Participants will be randomly assigned into two groups (n=15 each) via simple randomization.

The intervention group will undergo IMT using the POWERbreathe Plus device, 5 days per week for 4 weeks. Training will begin at 50% of the participants' MIP and increase by 10% each week, reaching 80% by the final week.

The control group will receive placebo IMT at a constant load equivalent to 15% of baseline MIP, following the same training schedule.

All interventions will be delivered in addition to the athletes' regular training programs. Pre- and post-intervention assessments will be conducted by a blinded physiotherapist who is not involved in the implementation of the training.

Assessment Parameters and Instruments To comprehensively evaluate the impact of IMT, objective and validated tools will be employed. Pulmonary function will be assessed using the Cosmed Pony FX device, measuring MIP, MEP, FEV1, FVC, and the FEV1/FVC ratio. Trunk endurance will be evaluated using the McGill Core Endurance protocol, which includes tests for trunk flexion, extension, and lateral plank. Muscle strength will be measured using the Isomed 2000 isokinetic dynamometer at a velocity of 60°/s to determine peak torque during trunk flexion and extension. Balance performance will be assessed with both the Y Balance Test (in anterior, posterolateral, and posteromedial directions) and the Flamingo Balance Test, which measures the ability to maintain single-leg stance. In addition, a participant tracking form will be used to record demographic information, training history, and attendance. All assessments will be performed under standardized conditions by a blinded evaluator.

Statistical Methods Appropriate statistical methods will be employed to analyze the data. Distribution characteristics and group comparisons will be assessed accordingly. Intra-group and inter-group differences, as well as time-by-group interactions, will be analyzed. Effect sizes will be calculated using standard procedures, and statistical significance will be set at p < 0.05.

Original Contribution of the Study This study is unique in its comprehensive evaluation of the effects of IMT not only on performance-related physical parameters but also on cardiopulmonary capacity in elite athletes. By focusing specifically on female wrestlers, the study contributes to sex-specific physiological research and is expected to provide evidence for the development of clinically applicable IMT protocols aimed at enhancing athletic performance and health.

ELIGIBILITY:
Inclusion Criteria:

1. To be an athlete in the Freestyle Women's Wrestling branch.
2. Participating in regular training at least 4 days a week.
3. To volunteer to participate in the study.
4. Being an athlete within TOHM for at least one year.
5. To be between the ages of 16-22.

Exclusion Criteria:

1. Have a cardiopulmonary disease that precludes the use of Pulmonary Function Testing.
2. Have specific balance problems (e.g., vestibular or neurological impairment).

Ages: 16 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal Inspiratory Pressure (MIP) [cmH₂O] | Baseline (Week 0) and Post-intervention (Week 4)
  Maximal inspiratory pressure (MIP) will be measured using the Cosmed Pony FX device. This value reflects the strength of inspiratory muscles before and after the intervention.
Change in Maximal Expiratory Pressure (MEP) [cmH₂O] | Baseline (Week 0) and Post-intervention (Week 4)
  Maximal expiratory pressure (MEP) will be assessed using the Cosmed Pony FX spirometer. It indicates the force generated by expiratory muscles and will be compared pre- and post-training.
Change in Forced Expiratory Volume in 1 Second (FEV1) [liters] | Baseline (Week 0) and Post-intervention (Week 4)
  FEV1 will be measured using the Cosmed Pony FX to evaluate pulmonary function. The value reflects the volume of air expelled in the first second of a forced exhalation.
Change in Forced Vital Capacity (FVC) [liters] | Baseline (Week 0) and Post-intervention (Week 4)
  FVC will be assessed with the Cosmed Pony FX device. It measures the total volume of air forcibly exhaled after a full inspiration, used to evaluate lung capacity changes due to training.
Change in FEV1/FVC Ratio [%] | Baseline (Week 0) and Post-intervention (Week 4)
  The FEV1/FVC ratio will be calculated from pulmonary function testing to assess airway function and efficiency. The ratio will be compared between baseline and after the 4-week intervention.

SECONDARY OUTCOMES:
Time Held in Trunk Flexion Test [seconds] | Baseline (Week 0) and Post-intervention (Week 4)
  Trunk flexion endurance will be assessed using the McGill Core Endurance Test Battery. The participant will maintain a trunk flexion position at a standardized angle. Duration will be recorded in seconds.
Time Held in Side Plank Test [seconds] | Baseline (Week 0) and post-intervention (Week 4)
  Lateral trunk endurance will be evaluated via the McGill side bridge (side plank) test. The time the participant can hold the position on each side will be recorded in seconds.
Time Held in Trunk Extension Test [seconds] | Baseline (Week 0) and Post-intervention (Week 4)
  Trunk extension endurance will be measured with the McGill Core Endurance Test Battery. The participant will hold the trunk in an extended position; the time maintained will be recorded in seconds.
Peak Torque of Trunk Flexors [Nm] | Baseline (Week 0) and Post-intervention (Week 4)
  Measured using the Isomed 2000 isokinetic dynamometer at 60°/s. Participants perform three trunk flexion repetitions; the highest peak torque value in Nm is recorded.
Peak Torque of Trunk Extensors [Nm] | Baseline (Week 0) and Post-intervention (Week 4)
  Measured using the Isomed 2000 isokinetic dynamometer at 60°/s. Participants perform three trunk extension repetitions; the highest peak torque in Nm is recorded.
Reach Distance in Y Balance Test - Anterior Direction [cm] | Baseline (Week 0) and Post-intervention (Week 4)
  The Y Balance Test will be used to assess dynamic balance. The maximum reach distance in the anterior direction will be measured in centimeters.
Reach Distance in Y Balance Test - Posteromedial Direction [cm] | Baseline (Week 0) and Post-intervention (Week 4)
  The Y Balance Test will be used to assess dynamic balance. The maximum reach distance in the posteromedial direction will be measured in centimeters.
Reach Distance in Y Balance Test - Posterolateral Direction [cm] | Baseline (Week 0) and Post-intervention (Week 4)
  The Y Balance Test will be used to assess dynamic balance. The maximum reach distance in the posterolateral direction will be measured in centimeters.
Time Maintained in Flamingo Balance Test [seconds] | Baseline (Week 0) and Post-intervention (Week 4)
  Static balance will be assessed using the Flamingo Balance Test. The time (in seconds) the participant can maintain a single-leg stance on a beam without losing balance will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs Üniversitesi, Samsun, Turkey (Türkiye)